CLINICAL TRIAL: NCT07310459
Title: Evaluation of Perinatal Risk Factors in Future Gross Motor Development of Preterm Infants: a Cross-sectional Study
Brief Title: Perinatal Risk Factors in Motor Development
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier Fernandez Rego, Doctor, Universidad de Murcia
Other Study IDs: CDIAT Lorca 1/2025
Record Dates: First submitted 2025-04-22; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Premature Infant; Risk Factors; Motor Development of Premature Infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of Preterm infants: Preterm infants cared at the "Fina Navarro Lopez" Childhood Development and Early Intervention Center (Lorca) between 2023 and 2025 who have been assessed using the Alberta Infant Motor Scale and the Perinatal Risk Inventory

SUMMARY:
The aim of this study is to analyze the effect of preterm gestational age, birth weight and perinatal risks factors on gross motor development of preterm infants.

We will compare the data of infants evaluated by the Alberta Infant Motor Scale (AIMS) and the Perinatal Risk Inventory (PERI) in an Infant Development and Early Intervention Center (IDEIC).

DETAILED DESCRIPTION:
An assessment of the infants' gross motor development will be carried out at admission, of IDEIC following the AIMS scale and bearing in mind their corrected age. Importantly, the trimester according to their corrected age was also recorded.

The gestational age of each infant will be recorded and used to group participants according to the following classification: late preterm newborn infant (LPNI; born between 34+1 and 36+6 weeks of gestation); moderate preterm newborn infant (MPNI; born between 32+1 to 34 weeks of gestation); very preterm newborn infant (VPNI; born between 28 to 32 weeks of gestation); and extreme preterm newborn infant (EPNI; born before 28 weeks of gestation).

The birth weight will be recorded and the infants will be grouped according to the following classification: newborns with adequate birth (birth weight of >2500 g), low birth weight (LBW; <2500 g and >1500 g); very low birth weight (VLBW; <2500 g and >1000 g), and extreme low birth weight (ELBW; <1000 g).

The infants will be assessed by the PERI test accounting for their discharge medical records. The infants will be then classified according to the biological risk level, in low, moderate and high risk.

Both the PERI and the AIMS test were assessed by three physiotherapists from the IDEIC with 10 to 20 years of experience.

Afterwards data will be analyzed using the Statistical Package for the Social Sciences Statistics (IBM SPSS) software for Windows version 22.0.

From all data collected as described in the brief summary, descriptive analysis and correlations between variables will be performed.

Samples will be classified using descriptive and frequency analysis. One-factor ANOVA, bivariate correlations will be carried out. Correlations between variables will be evaluated using Pearson's coefficient (bivariate correlation) or Spearman's coefficient (rank correlation). Frequencies analysis, square Chi test and backwards regression analysis will be used when appropriate.

AIMS direct scores will be standardized by converting them into Z scores. AIMS standard mean and deviation by age and gender will be used.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants showing biological risk factors
* parents or tutors signe an informed consent.

Exclusion Criteria:

* Diagnosis of encephalopathy
* genetic syndromes
* congenital malformations
* neuromuscular disorders
* myopathies
* metabolic and oncologic diseases

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The sample will consist of preterm infants referred to the IDEIC from the Neonatal Service of the Virgen de la Arrixaca University Hospital in Murcia, the Pediatrics Service of the Rafael Méndez University Hospital in Lorca, the Pediatric Service of Health Centers in Lorca area and/or by family referral.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal Risk Inventory (PERI) | Day 1
  The PERI is a test designed to assess neonatal situation, prior to infants' discharge from the hospital at birth that determines the possibility of abnormalities or pathologies in the infant' development at very early stages. Its predictive value is greater when it reaches a score equal or superior to 10.
  The infants will be assessed by the PERI test accounting using their discharge medical records.
Alberta Infant Motor Scale (AIMS) | Baseline
  The Alberta Infant Motor Scale (AIMS) is an observational scale to assess infants' gross motor development from birth to independent walking. The test consists of 58 items based on descriptions of the postural control in supine (9 items), prone (21 items), sitting (12 items) and standing (16 items) position. Each item scores one point, therefore the maximum puntuation possible is 58 points and the minimum 0 points. The greater the puntuation, the better is their motor development.
  It is conceived for infants from 0 to 18 months old. The test provides information about the infant's motor activities and allows the measurement of motor activity development over time or before and after therapy. The infants' assessment needs to take place in a quiet environment with minimal handling and without stimuli or random help. An assessment of the infants' gross motor development will be carried out at admission, following the AIMS scale and bearing in mind their corrected age.
Gestational age | Day 1
  Gestational age at birth. This information will be extracted from their discharge medical records
Birth weight | Day 1
  Weight that preterm infant had at birth. This information will be extracted from their discharge medical records

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Fernandez Rego, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- CDIAT Fina Navarro Lopez, Lorca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared upon justified request to the authors.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: indefinitely from the publication of the study
Access Criteria: Proper request to the authors.

REFERENCES:
- [Background] Pritchard MA, Colditz PB, Cartwright D, Gray PH, Tudehope D, Beller E. Risk determinants in early intervention use during the first postnatal year in children born very preterm. BMC Pediatr. 2013 Dec 5;13:201. doi: 10.1186/1471-2431-13-201. PMID 24304976
- [Background] Zaramella P, Freato F, Milan A, Grisafi D, Vianello A, Chiandetti L. Comparison between the perinatal risk inventory and the nursery neurobiological risk score for predicting development in high-risk newborn infants. Early Hum Dev. 2008 May;84(5):311-7. doi: 10.1016/j.earlhumdev.2007.08.003. Epub 2007 Sep 27. PMID 17897797
- [Background] Thomaidis L, Zantopoulos GZ, Fouzas S, Mantagou L, Bakoula C, Konstantopoulos A. Predictors of severity and outcome of global developmental delay without definitive etiologic yield: a prospective observational study. BMC Pediatr. 2014 Feb 12;14:40. doi: 10.1186/1471-2431-14-40. PMID 24521451
- [Background] Christian P, Murray-Kolb LE, Tielsch JM, Katz J, LeClerq SC, Khatry SK. Associations between preterm birth, small-for-gestational age, and neonatal morbidity and cognitive function among school-age children in Nepal. BMC Pediatr. 2014 Feb 27;14:58. doi: 10.1186/1471-2431-14-58. PMID 24575933